CLINICAL TRIAL: NCT04057118
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Dose Study to Evaluate the Efficacy and Safety of Oral SKI-O-703 in Patients With Active Rheumatoid Arthritis Despite Treatment With Conventional Therapies
Brief Title: A Study to Evaluate the Effectiveness and Safety of SKI-O-703 in Patients Experiencing Active Rheumatoid Arthritis Despite Treatment With Conventional Therapies.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oscotec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OSCO-P2201
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — cevidoplenib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SKI-O-703 100 mg (Experimental)
  Interventions: Drug: SKI-O-703
- SKI-O-703 200 mg (Experimental)
  Interventions: Drug: SKI-O-703
- SKI-O-703 400 mg (Experimental)
  Interventions: Drug: SKI-O-703
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SKI-O-703 — Oral administration, twice per day
  Arms: SKI-O-703 100 mg; SKI-O-703 200 mg; SKI-O-703 400 mg
Drug: Placebo — Oral administration, twice per day
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of SKI-O-703 compared with placebo, in patients with active rheumatoid arthritis (RA) who have had an inadequate response to conventional synthetic disease-modifying agents. Patients will be randomly assigned to one of 4 groups and will receive one of three doses of SKI-O-703 or placebo, administered orally twice daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide written, signed, informed consent.
* Patients must have a diagnosis of Rheumatoid Arthritis (RA) according to American College of Rheumatology (ACR) criteria or the 2010 ACR/European League Against Rheumatism classification, for at least 6 months prior to first administration of study drug.
* Patients must have active RA at screening and baseline (Day 1 of the study).
* Patients who have active disease despite csDMARD (conventional synthetic disease-modifying antirheumatic drugs) therapy for at least 3 months prior to Day 1 of the study.
* Patients must have had an inadequate response to previous anti-TNF⍺ (anti-tumor necrosis factor alpha) biological agent(s) for the treatment of RA and meet the washout period prior to Day 1 of the study.

Exclusion Criteria:

* Patients receiving oral agents, except for medications listed in inclusion criteria for the treatment of RA.
* Patients who have previously received any other or biological agent for the treatment of RA, other than anti-TNF⍺ inhibitor(s).
* Patients who have a current or past history of hepatitis B virus (HBV) infection; positive test for hepatitis C virus (HCV) antibody; positive test for human immunodeficiency virus (HIV); history of or concurrent interstitial pneumonia; acute infection requiring oral antibiotics within 2 weeks, or parenteral injection of antibiotics within 4 weeks prior to first administration of the study drug; other serious infection within 6 months prior to first administration of study drug; recurrent herpes zoster or other chronic or recurrent infection within 6 weeks prior to first administration of the study drug; past or current granulomatous infections or other severe or chronic infection; positive test for tuberculosis (TB) or other evidence of TB.
* Patients with uncontrolled diabetes mellitus, or uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg).
* Patients with any other inflammatory or rheumatic diseases that could impact the evaluation of the effect of the study drug.
* Patients with a history of malignancy within 5 years prior to first administration of the study drug, except completely excised and cured squamous cell carcinoma, carcinoma of the cervix in situ, cutaneous basal cell carcinoma, or cutaneous squamous cell carcinoma.
* New York Heart Association (NYHA) class III or IV heart failure, severe uncontrolled cardiac disease or heart attack within 6 months prior to first administration of the study drug.
* Female patients who are currently pregnant, breastfeeding or planning to become pregnant or breastfeed within 6 months of the last dose of the study drug.

Other protocol-defined inclusion/exclusion criteria could apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (12):
  - Oscotec Investigational Site (Site 3110), Beverly Hills, California
  - Oscotec Investigational Site (Site 3105), Upland, California
  - Oscotec Investigational (Site 3104), Miami Lakes, Florida
  - Oscotec Investigational Site (Site 3112), Tampa, Florida
  - Oscotec Investigational Site (Site 3108), Lexington, Kentucky
  - Oscotec Investigational Site (Site 3102), Oklahoma City, Oklahoma
  - Oscotec Investigational Site (Site 3107), Duncansville, Pennsylvania
  - Oscotec Investigational Site (3106), Carrollton, Texas
  - Oscotec Investigational Site (Site 3111), Houston, Texas
  - Oscotec Investigational Site (Site 3109), Mesquite, Texas
  - Oscotec Investigational Site (Site 3103), San Antonio, Texas
  - Oscotec Investigational Site (Site 3101), Tomball, Texas
- Czechia (2):
  - Oscotec Investigational Site (Site 2101), Ostrava
  - Oscotec Investigational Site (Site 2102), Zlín
- Poland (8):
  - Oscotec Investigational Site (Site 2203), Poznan, Greater Poland Voivodeship
  - Oscotec Investigational Site (Site 2204), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Oscotec Investigational Site (Site 2208), Wroclaw, Lower Silesian Voivodeship
  - Oscotec Investigational Site (Site 2207), Lublin, Lublin Voivodeship
  - Oscotec Investigational Site (Site 2202), Warsaw, Masovian Voivodeship
  - Oscotec Investigational Site (Site 2201), Bialystok, Podlaskie Voivodeship
  - Oscotec Investigational Site (Site 2206), Nadarzyn
  - Oscotec Investigational Site (Site 2209), Ostrowiec Świętokrzyski, Świętokrzyskie Voivodeship
- Russia (8):
  - Oscotec Investigational Site (Site 2307), Kemerovo
  - Oscotec Investigational Site (Site 2304), Moscow
  - Oscotec Investigational Site (Site 2305), Moscow
  - Oscotec Investigational Site (Site 2308), Novosibirsk
  - Oscotec Investigational Site (Site 2306), Ryazan
  - Oscotec Investigational Site (Site 2302), Saint Petersburg
  - Oscotec Investigational Site (Site 2303), Saint Petersburg
  - Oscotec Investigational Site (Site 2301), Tomsk
- Ukraine (10):
  - Oscotec Investigational Site (Site 2510), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Oscotec Investigational Site (Site 2505), Ternopil, Ternopil Oblast
  - Oscotec Investigational Site (Site 2506), Vinnytsia, Vinnytsia Oblast
  - Oscotec Investigational Site (Site 2504), Vinnytsia, Vinnytsia Oblast
  - Oscotec Investigational Site (Site 2508), Kharkiv
  - Oscotec Investigational Site (Site 2501), Kyiv
  - Oscotec Investigational Site (Site 2503), Kyiv
  - Oscotec Investigational Site (Site 2502), Kyiv
  - Oscotec Investigational Site (Site 2507), Poltava
  - Oscotec Investigational Site (Site 2509), Vinnytsia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | SKI-O-703 100 mg | SKI-O-703 200 mg | SKI-O-703 400 mg
Started | 41 | 41 | 40 | 41
Completed | 38 | 39 | 37 | 36
Not Completed | 3 | 2 | 3 | 5
Not completed — Adverse Event | 1 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 2
Not completed — Not Specific | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | SKI-O-703 100 mg | SKI-O-703 200 mg | SKI-O-703 400 mg | Total
Number analyzed (Participants) | 41 | 41 | 40 | 41 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (12.03) | 56.8 (10.90) | 55.2 (11.51) | 52.3 (12.80) | 54.9 (11.84)
Age, Customized [Count of Participants; unit: Participants]
  Age Category: Less than 65 years old | 30 | 31 | 31 | 36 | 128
  Age Category: Greater than 65 to less than 75 years old | 9 | 9 | 9 | 3 | 30
  Age Category: 75 years old or greater | 2 | 1 | 0 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 29 | 32 | 33 | 128
  Male | 7 | 12 | 8 | 8 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 36 | 41 | 37 | 38 | 152
  Race: Black or African-American | 3 | 0 | 1 | 0 | 4
  Race: Asian | 2 | 0 | 0 | 2 | 4
  Race: American-Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Race: Other | 0 | 0 | 2 | 0 | 2
Height (cm) [Mean (Standard Deviation); unit: centimeter] | 166.07 (5.995) | 165.61 (9.003) | 163.33 (7.918) | 163.18 (8.098) | 164.55 (7.867)
Weight (kg) [Mean (Standard Deviation); unit: kilogram] | 75.68 (12.590) | 77.09 (16.243) | 78.71 (20.177) | 70.83 (13.372) | 75.56 (15.973)
Body mass index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 27.48 (4.602) | 28.04 (5.076) | 29.50 (7.474) | 26.56 (4.357) | 27.88 (5.555)
Time since RA onset (years) [Mean (Standard Deviation); unit: years] | 9.05 (6.418) | 6.86 (5.587) | 6.12 (5.578) | 8.83 (7.260) | 7.72 (6.321)
Nicotine use [Count of Participants; unit: Participants]
  Never a smoker or user | 34 | 32 | 30 | 31 | 127
  Prior smoker or user | 2 | 4 | 6 | 2 | 14
  Current smoker or user | 5 | 5 | 4 | 8 | 22
Alcohol history [Count of Participants; unit: Participants]
  Never a drinker | 32 | 34 | 27 | 31 | 124
  Prior drinker, but no longer a drinker | 2 | 3 | 2 | 2 | 9
  Current drinker | 7 | 4 | 11 | 8 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Disease Activity Score
Description: Mean change from baseline in disease activity score for 28 joints (DAS28) using hsCRP (high sensitivity C-reactive protein).
  Disease Activity Score (DAS) modified to include 28 joint count (DAS28) consisted of composite score of following variables: tender joint count (TJC28), swollen joint count (SJC28), and high sensitivity C-reactive protein (hsCRP) (milligrams per liter). DAS28 was calculated using following formula: DAS28-CRP=0.56*square root (sqrt)(TJC28)+0.28*sqrt(SJC28)+0.36*natural log(hsCRP+1)*1.10+1.15.
  High DAS28-hsCRP value indicates more severe disease activity, by value of >5.1 indicating relatively high disease activity, whereas value of <3.2 indicating achieved lower disease activity (no theoretical full range available).
Time Frame: Baseline and Week 12
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SKI-O-703 100 mg | SKI-O-703 200 mg | SKI-O-703 400 mg
Number analyzed (Participants) | 37 | 36 | 36 | 36
score on a scale | -0.95 (0.152) | -0.91 (0.155) | -1.06 (0.155) | -1.15 (0.155)

2. Secondary Outcome: • Percentage of Patients With ACR20 (American College of Rheumatology 20) Score
Description: ACR20 score is the percentage of patients showing ≥20% improvement from baseline in tender joint count (68 joint counts), ≥20% improvement in swollen joint count (66 joint counts), and ≥20% improvement in at least 3 of the following: patient's global assessment of arthritis pain; patient's global assessment of disease activity; physician's global assessment of disease activity; health assessment questionnaire-disability index (HAQ-DI); hsCRP (high sensitivity C-reactive protein)
Time Frame: Baseline and Weeks 2, 4 8 and 12
Population: The number analyzed in some rows decreased as weeks increased, as some patients withdrew from the study or had missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SKI-O-703 100 mg | SKI-O-703 200 mg | SKI-O-703 400 mg
Number analyzed (Participants) | 27 | 29 | 28 | 24
Participants
  Week 2 | 2 | 3 | 5 | 5
  Week 4: number analyzed (Participants) | 27 | 29 | 27 | 24
  Week 4 | 7 | 4 | 6 | 9
  Week 8: number analyzed (Participants) | 26 | 29 | 26 | 22
  Week 8 | 10 | 9 | 9 | 7
  Week 12: number analyzed (Participants) | 25 | 26 | 25 | 21
  Week 12 | 12 | 9 | 14 | 9

3. Secondary Outcome: • Percentage of Patients With ACR50 (American College of Rheumatology 50) Score
Description: ACR50 score is the percentage of patients showing ≥50% improvement from baseline in tender joint count (68 joint counts), ≥50% improvement in swollen joint count (66 joint counts), and ≥50% improvement in at least 3 of the following: patient's global assessment of arthritis pain; patient's global assessment of disease activity; physician's global assessment of disease activity; health assessment questionnaire-disability index (HAQ-DI); hsCRP (high sensitivity C-reactive protein)
Time Frame: Baseline and Weeks 2, 4 8 and 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SKI-O-703 100 mg | SKI-O-703 200 mg | SKI-O-703 400 mg
Number analyzed (Participants) | 27 | 29 | 28 | 24
Participants
  Week 2 | 0 | 0 | 0 | 2
  Week 4: number analyzed (Participants) | 27 | 29 | 27 | 24
  Week 4 | 2 | 2 | 1 | 6
  Week 8: number analyzed (Participants) | 25 | 29 | 26 | 22
  Week 8 | 3 | 4 | 4 | 5
  Week 12: number analyzed (Participants) | 25 | 26 | 25 | 21
  Week 12 | 4 | 4 | 6 | 5

4. Secondary Outcome: • Percentage of Patients With ACR70 (American College of Rheumatology 70) Score
Description: ACR70 score is the percentage of patients showing ≥70% improvement from baseline in tender joint count (68 joint counts), ≥70% improvement in swollen joint count (66 joint counts), and ≥70% improvement in at least 3 of the following: patient's global assessment of arthritis pain; patient's global assessment of disease activity; physician's global assessment of disease activity; health assessment questionnaire-disability index (HAQ-DI); hsCRP (high sensitivity C-reactive protein)
Time Frame: Baseline and Weeks 2, 4 8 and 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SKI-O-703 100 mg | SKI-O-703 200 mg | SKI-O-703 400 mg
Number analyzed (Participants) | 27 | 29 | 28 | 24
Participants
  Week 2 | 0 | 0 | 0 | 1
  Week 4: number analyzed (Participants) | 27 | 29 | 27 | 24
  Week 4 | 0 | 0 | 0 | 1
  Week 8: number analyzed (Participants) | 26 | 29 | 26 | 22
  Week 8 | 0 | 0 | 2 | 3
  Week 12: number analyzed (Participants) | 25 | 26 | 25 | 21
  Week 12 | 1 | 0 | 3 | 3

5. Secondary Outcome: Health Assessment Questionnaire-Disability Index (HAQ-DI) Score
Description: Change from baseline measured by disability index
  The Health Assessment Questionnaire-Disability Index (HAQ-DI) is a subject-reported questionnaire that is commonly used to measure the disease associated disability. It consists of 8 sections which are dressing or grooming, arising, eating, walking, hygiene, reaching, gripping, and performing other daily activities.
  Scores for each functional area were averaged to calculate HAQ-DI scores, ranging from 0 (no disability) to 3 (worst disability), higher score showing more disability.
  A decrease in HAQ-DI score indicated an improvement in the participant's condition.
Time Frame: Baseline and Weeks 2, 4 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | SKI-O-703 100 mg | SKI-O-703 200 mg | SKI-O-703 400 mg
Number analyzed (Participants) | 41 | 41 | 40 | 41
score on a scale
  Change from Baseline at Week 2: number analyzed (Participants) | 40 | 40 | 39 | 39
  Change from Baseline at Week 2 | -0.0969 (0.3171) | -0.1375 (0.2953) | -0.2340 (0.3037) | -0.3397 (0.4035)
  Change from Baseline at Week 4: number analyzed (Participants) | 39 | 40 | 38 | 39
  Change from Baseline at Week 4 | -0.2179 (0.3228) | -0.2906 (0.3494) | -0.2895 (0.2979) | -0.3718 (0.4646)
  Change from Baseline at Week 8: number analyzed (Participants) | 38 | 40 | 37 | 36
  Change from Baseline at Week 8 | -0.3816 (0.4171) | -0.3781 (0.3968) | -0.3311 (0.4362) | -0.4306 (0.5040)
  Change from Baseline at Week 12: number analyzed (Participants) | 37 | 36 | 36 | 36
  Change from Baseline at Week 12 | -0.4459 (0.4765) | -0.5208 (0.4758) | -0.4444 (0.5040) | -0.4514 (0.5246)

6. Secondary Outcome: Adverse Events (AEs)
Time Frame: Up to Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SKI-O-703 100 mg | SKI-O-703 200 mg | SKI-O-703 400 mg
Number analyzed (Participants) | 41 | 41 | 40 | 41
Participants
  Participants with any Treatment Emergent Adverse Event (TEAE) | 19 | 16 | 23 | 25
  Participants with any treatment-related TEAE | 8 | 4 | 12 | 14

7. Secondary Outcome: Serious Adverse Events (SAEs)
Time Frame: Up to Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SKI-O-703 100 mg | SKI-O-703 200 mg | SKI-O-703 400 mg
Number analyzed (Participants) | 41 | 41 | 40 | 41
Participants
  Participants with any treatment-emergent SAE | 1 | 1 | 0 | 1
  Participants with any treatment-related, treatment-emergent SAE | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: At every study visit, subjects were asked a standard nonleading question to explore a response regarding any medically related changes in their well-being. They were also asked if they had been hospitalized or had any accidents. In addition to subject observations, AEs identified from any study data (eg, laboratory values, physical examination findings, ECG changes) or identified from review of other documents that were relevant to subject safety were documented.
Arm/Group | Placebo | SKI-O-703 100 mg | SKI-O-703 200 mg | SKI-O-703 400 mg
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41 | 0/40 | 0/41
Serious Adverse Events (participants affected / at risk) | 1/41 | 1/41 | 0/40 | 1/41
Other Adverse Events (participants affected / at risk) | 8/41 | 6/41 | 10/40 | 13/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | SKI-O-703 100 mg (N=41) | SKI-O-703 200 mg (N=40) | SKI-O-703 400 mg (N=41)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Myocarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | SKI-O-703 100 mg (N=41) | SKI-O-703 200 mg (N=40) | SKI-O-703 400 mg (N=41)
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 3
Headache (Nervous system disorders) | 2 | 1 | 6 | 6
Nausea (Gastrointestinal disorders) | 2 | 0 | 3 | 2
Constipation (Gastrointestinal disorders) | 4 | 3 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT04057118/Prot_002.pdf
  • Statistical Analysis Plan (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT04057118/SAP_001.pdf